CLINICAL TRIAL: NCT06655714
Title: Evaluation of Inadequate Response to Ultrasound-Guided Subacromial Corticosteroid Injection in Shoulder Impingement Syndrome: Treatment Failure or Central Sensitization?
Brief Title: Evaluation of Inadequate Response to Ultrasound-Guided Subacromial Corticosteroid Injection in Shoulder Impingement Syndrome
Status: Completed | Type: Observational
Sponsor: Beylikduzu State Hospital (Other)
Responsible Party: Principal Investigator, Busra Sirin, Principle Investigator, Beylikduzu State Hospital
Other Study IDs: BeylikduzuStateH7
Record Dates: First submitted 2024-10-22; First posted 2024-10-23 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Impingement Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with adequate response: In this study, patients whose Visual Analog Scale (VAS) score decreases by 50% or more after 4 weeks of receiving the ultrasound-guided corticosteroid injection will be considered to have had an adequate response.
  Interventions: Other: No intervention
- Patients with inadequate response: In this study, an inadequate response is defined as less than a 50% reduction in pain, as measured by the Visual Analog Scale (VAS), four weeks after the ultrasound-guided corticosteroid injection.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The aim of this study is to investigate the impact of central sensitization in patients with shoulder impingement syndrome who have shown an inadequate response to ultrasound-guided subacromial corticosteroid injection. Additionally, the patients' pain perception and emotional state will be evaluated, and the relationships between these factors and the treatment response will be analyzed.

DETAILED DESCRIPTION:
Seventy-two patients aged 18-75, who applied to the Physical Therapy and Rehabilitation outpatient clinic at Beylikdüzü State Hospital, diagnosed with shoulder impingement syndrome based on magnetic resonance imaging (MRI), and who received ultrasound-guided corticosteroid injection, will be included in the study. No additional interventions or procedures will be performed for the research. These patients, who were previously assessed and treated in the outpatient clinic, will be invited for a follow-up examination at the 4th week after the injection. During the follow-up, their response to the treatment will be evaluated using the Visual Analog Scale (VAS). A reduction of less than 50% on the VAS by the end of the 4th week will be considered an inadequate response. Patients with inadequate and good responses will be divided into two groups and assessed for central sensitization, pain perception, and emotional state. Central sensitization will be evaluated using the Central Sensitization Inventory (CSI), and hyperalgesia will be assessed using an algometer to measure pressure-pain threshold. Additionally, the Pain Catastrophizing Scale and the Hospital Anxiety and Depression Scale will be used to determine the patients' emotional state and pain perception.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65.
* Diagnosed with shoulder impingement syndrome.
* Received ultrasound-guided subacromial corticosteroid injection.
* Experienced shoulder pain for at least 6 months.

Exclusion Criteria:

* History of surgery or fracture in the shoulder or related areas.
* Presence of an active infection.
* Received shoulder injection within the last 6 months.
* Underwent physical therapy for the shoulder in the last 6 months.
* Presence of other musculoskeletal or neurological conditions that could cause shoulder pain (e.g., cervical disc herniation, stenosis, moderate to severe osteoarthritis, adhesive capsulitis, rheumatologic pathologies, infectious joint diseases).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include 72 patients aged 18-65 who have been diagnosed with shoulder impingement syndrome and have undergone ultrasound-guided subacromial corticosteroid injection.
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 0 day, 4th week
  The Visual Analog Scale is a tool used to measure the intensity of pain. It consists of a 10 cm line, where one end represents "no pain" (0) and the other end represents "worst imaginable pain" (10). Patients mark the point on the line that reflects their current pain level. In this study, a reduction of less than 50% on the VAS after 4 weeks is considered an inadequate response to the treatment.
Central Sensitization Inventory (CSI) | 0 day, 4th week
  The CSI is a self-reported questionnaire used to identify the presence of central sensitization, which is a condition where the central nervous system becomes hypersensitive to stimuli. It consists of 25 items that measure symptoms related to central sensitization syndromes. Higher scores indicate a greater likelihood of central sensitization, which can contribute to persistent pain in conditions like shoulder impingement syndrome.
Pressure-Pain Threshold (PPT) Using Algometer | 0 day, 4th week
  The Pressure-Pain Threshold is the minimum force applied to the skin that induces pain. In this study, an algometer is used to measure PPT at various points on the body. Lower PPT values indicate increased sensitivity to pressure, which is a sign of hyperalgesia, often associated with central sensitization.
Pain Catastrophizing Scale (PCS): | 0 day, 4th week
  The PCS is a psychological tool used to assess the extent to which individuals experience catastrophic thoughts related to their pain. It includes 13 items that measure rumination, magnification, and helplessness in response to pain. Higher scores on the PCS suggest that the patient tends to catastrophize pain, which can negatively affect their pain experience and recovery.
Hospital Anxiety and Depression Scale (HADS): | 0 day, 4th week
  The HADS is a questionnaire used to assess the emotional state of patients, focusing on anxiety and depression. It consists of 14 items, divided into two subscales: one for anxiety (HADS-A) and one for depression (HADS-D). Higher scores indicate greater levels of anxiety or depression, which can influence how patients perceive and cope with their pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Beylikdüzü State Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sirin Ahisha B, Paker N, Kesiktas N, Bugdayci ND, Ahisha YC. Evaluation of Inadequate Response to Ultrasound-Guided Subacromial Corticosteroid Injection in Shoulder Impingement Syndrome: Treatment Failure or Central Sensitization? Arch Phys Med Rehabil. 2025 Aug;106(8):1227-1237. doi: 10.1016/j.apmr.2025.01.469. Epub 2025 Feb 1. PMID 39900325